CLINICAL TRIAL: NCT04084743
Title: Concurrent Dual Task and Virtual Reality Innovation to Improve Balance, Posture and Gait in Patients With Parkinson Disease
Brief Title: Dual Task and Virtuality Training Innovation to Improve Balance, Posture and Gait in Patients With Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/2019/01; U1111-1234-9952 (Other: UTN by WHO International Critical Trial Registry Platform)
Record Dates: First submitted 2019-08-31; First posted 2019-09-10 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: Virtual reality; Targeted therapy; Computer game
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality training and Dual task intervention (Experimental): Cognitive and motor Dual-task intervention and virtual reality training intervention in patients with Parkinson's disease
  Interventions: Other: Virtual reality intervention; Other: Dual task intervention; Other: Conventional physiotherapy
- Conventional physiotherapy and Dual task intervention (Active Comparator): The dual-task intervention without virtual reality training intervention in patients with Parkinson's disease
  Interventions: Other: Virtual reality intervention; Other: Dual task intervention; Other: Conventional physiotherapy

INTERVENTIONS:
Other: Virtual reality intervention — Virtual reality intervention includes: Maze game software
Other: Dual task intervention — The intervention combined both motor and cognitive training which includes, walking 10 meter (1) Free walking (2) Walking carrying an emptying tray (3) Walking carrying a tray with 4 empty glasses (4) Digit calculations (Counting forward and backward, addition, subtraction, multiplication and division) during walking.
Other: Conventional physiotherapy — 1. Gait training in parallel bar
  2. Balance activities which includes, a. Forward direction activity b. Backward direction activity c. Sideways direction activity

SUMMARY:
Individuals affected with Parkinson disease (PD), are found to be at high risk of motor impairment and non-motor impairment as well. It further leads to affect the quality of life in patients of PD, due to impairments in postural instability, balance impairment and gait disturbances. Hence, various Physiotherapy based rehabilitation is on-demand that improves their quality of life and prognosis. Emerging trends in neuro-rehabilitation are Virtual reality intervention (VRI), that helps the patient to involve in a virtual environment and provide rehabilitation as per need by using different software games. As a result, their balance, posture and gait can improve speedily. In VRI we will be using the latest model of VRI that will include an assessment tool to assess the disability and provide rehabilitation. The cognitive system is also get affected due to physiological changes occur in PD, that leads to impair the other functions during walking such as balance and posture. Because during walking they can not perform dual task orientation to correct their posture and balance. So, dual-task intervention (DTI) is helpful to train them and involve them to participate actively in various activities.

In this project, we will develop an innovative rehabilitation technique to improve the posture, balance and gait in patients with PD. It will include VRI and additive DTI that will keep the patients motivated to perform the exercise actively. To assess the problems we will use standard device posturography that will be used before the intervention and after the intervention to identify the changes in their condition. Additionally, we will use some scales as outcome measures to assess the PD, quality of life and gait. Previous studies show that VR games and dual-task intervention training are an effective method to rehabilitate neurological ill patients. During the experiments, both conventional (DTI) and experimental (VRI+ DTI) will be considered.

DETAILED DESCRIPTION:
Introduction Parkinson disease (PD) is a neurodegenerative disease of the brain, leads to degeneration and causing the motor and non-motor symptoms. PD is characterized by dopaminergic neurotransmitter deficiency. It is a progressive neurological condition that affects more than 10 million people worldwide. Cardinal features of PD are bradykinesia, rigidity and tremor are common symptoms. But gait, postural instability and balance are common risk factors for falling in these population and have a great impact on the quality of life.

There are various treatments available in the pharmacological and surgical field. However, their effectiveness is not satisfying much and invasive procedures are not cost-effective. With the progression of disease patent often become less responsive to medication and develop various difficulties in their daily activities.

Therefore, Physiotherapy(PT) interventions are very important to rehabilitate the patients affected with PD. It helps to improve movement function, motor performance and increase the quality of life. There is active participation from the side of the patient will be there that keeps the patients motivated.

Among emerging approaches in the field of PT, virtual reality(VR) has been proposed as an innovative and effective method for improving gait, balance and postural instability. Patients of PD faces cognitive impairment which leads to impaired attention during their gait because they are unable to put attention on their posture and balance. So attention is responsible for maintaining posture and gait, leads to reduce dual-task ability which is very important in our daily life activities. So to improve the quality of life by correcting posture and gait cognitive dual-task intervention training plays important role in rehabilitation.

Various studies suggested single intervention to improve gait, posture and balance ability in PD patients. To our knowledge, no study investigated the possibility to apply VR with dual-task intervention. the current study compares the effects of VR intervention (VRI) and cognitive dual-task intervention(DTI) between posture, balance and gait. To our knowledge, this will be the first study to compare VRI and DTI on a variety of motor tasks in the homogenous group in their OFF period of medication state.

We hypothesized that addition of VRI with DTI can lead to improve the balance, postural instability and gait in patients with PD and can slow the progression of the disease without changing the medication plan.

2. Materials and Methods: Ethical statement and subject recruitment The study protocol was approved by the institutional research advisory committee (RAC) and registered under the Universal Trial Number (UTN). The protocol will be registered under ClinicalTrials.gov, under World Health Organization International Clinical Trials Registry Platform and then the study will be submitted for the ethical approval by the institutional ethics committee of Maharishi Markandeshwar Deemed to Be University, Mullana, Haryana with a unique reference number. The study will be executed in accordance with the principles of the Declaration of Helsinki (Revised, 2013) and National ethical guidelines for Biomedical and Health research involving human participants by Indian council for medical research (ICMR, 2017). The purpose of the study will be clearly explained to the patient with Parkinson disease. A written informed consent form will be obtained from the recruited patients.

Inclusion criteria Idiopathic PD (According to the united kingdom Parkinson's disease society brain bank criteria) Hoehn and Yahr stage III Able to walk without any assistance Age between45-70 Both sex male and female Exclusion criteria Any neurological disease other than PD Vestibular disorders Urinary incontinence Musculoskeletal impairments that could affect gait Inability to stand and walk unassisted Uncooperative patients Random Allocation Total of X patient with Parkinson disease was screened and through convenience sampling method, n patients were selected based on the inclusion criteria for the double, blind three-group pretest-posttest randomized controlled design. Demographic data will be recorded for all the patients. The patient with PD will be allocated in three groups, dual-task treatment group (DTG), virtual reality treatment group (VRG) and daily physiotherapy group (DPG) by compute generated block randomization technique. According to it, there will be n blocks, with the matrix design of n × N, where n being rowed. Each row could have n blocks, patients will be allotted to one of the three groups based on the randomly generated number by computer. Once all the first row will be allotted, then the next row block will be opened for enrolment. The advantage of this method of randomization is that the number of patients assigned to each group over time would have been approximately equal. By this, the unequal allocation of sample size will be avoided. The outcome assessor and the participants involved in the intervention will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD (according to the united kingdom parkinson's disease society brain bank criteria)
* Hoehn and Yahr stage III
* Able to walk without any assistance
* Age between 45-70
* Both sex male and female

Exclusion Criteria:

* Any neurological disease other than PD
* Vestibular disorders
* Musculoskeletal impairments that could affect gait
* Inability to stand and walk unassisted
* Uncooperative patients

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-06-02 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire | change will be measured at baseline and after 4 weeks of intervention
  It is a 39 item self report questionnaire, which assess Parkinson disease specific health related quality of the patients. It assess experienced difficulty impact of PD in functioning and well being.
Posturography | change will be measured at baseline and after 4 weeks of intervention
  BIORescue (system for sequential posture analysis and rehabilitation- made in France) allows carrying out a comparative assessment supported by many analyses repeated at different times throughout the treatment. Several types of exercises make it possible to work on the reestablishment of the transfer of the support, the stability, the balance, the anticipation of movement, etc.

SECONDARY OUTCOMES:
UPDRS | change will be measured at baseline and after 4 weeks of intervention
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's Disease in patients. The UPDRS scale consist of te following five segments: (1) Mentation, Behaviour, and Mood, (2) ADL ,(3) Motor section,(4) Modified Hoehn and Yahr scale, (5)Schwab and England ADL scale. Each answer to the scale is evaluated by a medical professional that specializes in Parkinson's disease during patient interviews. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh K Srivastav, MPT, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hubbard B, Pothier D, Hughes C, Rutka J. A portable, low-cost system for posturography: a platform for longitudinal balance telemetry. J Otolaryngol Head Neck Surg. 2012 Apr;41 Suppl 1:S31-5. PMID 22569047
- [Result] Abdolahi A, Scoglio N, Killoran A, Dorsey ER, Biglan KM. Potential reliability and validity of a modified version of the Unified Parkinson's Disease Rating Scale that could be administered remotely. Parkinsonism Relat Disord. 2013 Feb;19(2):218-21. doi: 10.1016/j.parkreldis.2012.10.008. Epub 2012 Oct 25. PMID 23102808
- [Result] Reinkensmeyer DJ, Boninger ML. Technologies and combination therapies for enhancing movement training for people with a disability. J Neuroeng Rehabil. 2012 Mar 30;9:17. doi: 10.1186/1743-0003-9-17. PMID 22463132
- [Result] Bisson E, Contant B, Sveistrup H, Lajoie Y. Functional balance and dual-task reaction times in older adults are improved by virtual reality and biofeedback training. Cyberpsychol Behav. 2007 Feb;10(1):16-23. doi: 10.1089/cpb.2006.9997. PMID 17305444
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22569047
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23102808
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22463132
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/17305444